CLINICAL TRIAL: NCT04682262
Title: The Effect of Cervical Dilatation on Pain in Nulliparous Women With Primary Dysmenorrhea.
Brief Title: The Effect of Cervical Dilatation on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Murat Yassa, Principal Investigator, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDPD
Record Dates: First submitted 2020-12-09; First posted 2020-12-23 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Dysmenorrhea Primary
Keywords: cervical dilatation; dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Labor Stage, First

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator diagnosed primary dysmenorrhea with clinical history and anamnesis. Investigator refers the patient to the surgical nurse and nurse performs the randomization process and prepare the patient (control group) for the cervical dilatation and hysteroscopy and schedule the control group for follow-up (expectant). The outcomes assessor is also blind to the assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical dilatation (Experimental): Patients receive cervical dilatation up to 10 millimeter Hegar dilator under general anaesthesia. Patient undergo standard hysteroscopy operation.
  Interventions: Procedure: Cervical dilatation
- Expectant (No Intervention): Patients are scheduled for follow-up.

INTERVENTIONS:
Procedure: Cervical dilatation — Patients undergo to cervical dilatation prior to the hysteroscopy under general anaesthesia with using Hegar dilator (no.10)
  Arms: Cervical dilatation

SUMMARY:
Primary dysmenorrhea (PD) is defined as recurrent, crampy pain occurring with menses in the absence of identifiable pelvic pathology. Standard initial management of PD includes NSAIDs as a first-line treatment and oral contraceptives for the relief of pain and improved daily activity. In patients who have persistent dysmenorrhea despite medical therapy of NSAIDs and/or oral contraceptives, further investigation including pelvic ultrasound, hysteroscopy or laparoscopy may be needed to rule out other underlying pathologies. Historically, It is an old clinical observation that primary dysmenorrhea is often completely or partially relieved by childbearing. Similarly, the investigators have observed that the diagnostic/operative hysteroscopy led to relive of pain in most of the cases in our practice. Therefore, the investigators hypothesized that the process of cervical dilatation can have a role in reducing pain of patients with dysmenorrhea. In this randomized, controlled study, it was aimed to assess the effect of operational cervical dilatation on the pain in patients with primary dysmenorrhea.

DETAILED DESCRIPTION:
Patients who applies to the outpatient clinic for reasons non-related to the dysmenorrhea (e.g. infertility investigation) will be assessed for the presence of primary dysmenorrhea by history taking and anamnesis. Patients will be randomized to have cervical dilatation and hysteroscopy or no intervention until the follow-up duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who applies to the outpatient clinic for reasons non-related to the dysmenorrhea (e.g. infertility investigation)
* Patients whose history and anamnesis indicate primary dysmenorrhea.
* Aged over 18 years old
* Nulliparous women

Exclusion Criteria:

* History of uterine surgery/operation
* History and clinical examinations which are indicative of secondary dysmenorrhea (Endometriosis, Adenomyosis, Uterine myomas, Endometrial polyps, Cervical stenosis, etc.)
* Positive pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-04-14 (Estimated); Study Completion 2021-05-21 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | Change between these periods: preoperative, postoperative 1st month, postoperative 2nd month
  Patients are asked to mark their pain on a 10 point visual scale which variate between 0 (no pain) to 10 (unbearable pain).
Verbal multidimensional scoring system for assessment of dysmenorrhea severity | Change between these periods: preoperative, postoperative 1st month, postoperative 2nd month
  This scale assess the dysmenorrhea by grading the severity. The assessment includes working ability, systemic symptoms and the use of analgesics. The grades vary between grade 0, grade 1 (mild), grade 2 (moderate) and grade 3 (severe).
EQ-5D | Change between these periods: preoperative, postoperative 1st month, postoperative 2nd month
  The EuroQol-5D (EQ-5D) is an instrument for measuring quality of life and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

OTHER OUTCOMES:
dyspareunia | Change between these periods: preoperative, postoperative 1st month, postoperative 2nd month
  Dyspareunia is assessed by a non-validated question if she feels disturbing pain during the sexual coitus or not (present / absent).

CONTACTS AND LOCATIONS:
Overall Officials: Niyazi Tug, MD, Prof, Study Director — Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Locations (1):
- Sehit Prof Dr Ilhan Varank Sancaktepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Upon request

REFERENCES:
- [Background] Gregersen H, Hee L, Liao D, Uldbjerg N. Distensibility and pain of the uterine cervix evaluated by novel techniques. Acta Obstet Gynecol Scand. 2016 Jul;95(7):717-23. doi: 10.1111/aogs.12891. Epub 2016 Mar 30. PMID 26946059